CLINICAL TRIAL: NCT02680873
Title: Efficacy of Single Anastomosis Sleeve Ileal (SASI) Bypass for Type-2 Diabetic Obese Patients: Loop Gastric Bipartition, a Novel Metabolic Surgery Procedure.
Brief Title: Efficacy of SASI Bypass for Type-2 Diabetic Obese Patients
Acronym: SASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, tarek mahdy, professor of surgery, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QASMSD5188453
Record Dates: First submitted 2016-02-07; First posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus Type 2 in Obese
Keywords: type 2 diabetes , obesity , SASI
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SASI bypass (Other): sleeve gastrectomy done and gastro-ileum anastomosis 2.5 meter from the ileocecal valve . the anastomosis is less than 3cmm in diameter . the concept to push undigested food early to the ileum to stimulate intestinal hormones secretion to control diabetes .
  Interventions: Other: SASI bypass

INTERVENTIONS:
Other: SASI bypass — he operation was done under general anesthesia. The technique commences with the devascularization of the greater curvature of the stomach with the harmonic scalpel.junction. The stomach is then tubularized over a 36 French calibration tube, with a linear stapler charged with a green cartridge, commencing 6 cm proximal to the pylorus. The ileocecal junction is identified and 250 cm is measured upwards. The selected loop is ascended antecolic without division of the greater omentum, and a stapled isoperistaltic side-to-side to the anterior wall of the antrum of the stomach just cranial 3 cm away from the pylorus with a linear stapler charged with a green cartridge.

SUMMARY:
the investigator modified the Sanator's operation by performing a loop rather than Roux-en-Y bipartition reconstruction and the investigator are reporting the first clinical results of the outcomes of SASI bypass as a mode of functional restrictive and neuroendocrine modulation therapeutic option for obese type 2 diabetes mellituspatients.

DETAILED DESCRIPTION:
All patients were subjected to thorough history, clinical examination and laboratory investigations including basic preoperative investigations, lipid profile, thyroid and suprarenal hormonal evaluation. In addition, patients may undergo further assessment for pulmonary functions or gastroesophageal disease including endoscope. . Abdominal ultrasound was done to exclude calcular cholecystitis and to evaluate the degree of fatty liver. Reduction the size of fatty liver was done by putting all patients on low-calorie protein diet for 6 weeks. Deep vein thrombosis prophylaxis started 12 h before surgery with low molecular weight heparin subcutaneous injections . Preoperative data included age, gender, initial weight, initial body mass index (BMI), obesity comorbidities and treatment medications used (chest problems, diabetes, arterial hypertension and cardiac ischaemia, hyperlipidemia, obstructive sleep apnea syndrome, gall stones, urinary stress incontinence, joint pain, depression, infertility and heart burn). Postoperative data included hospital stay, early postoperative complications during the first month (e.g. fever, collection, bleeding, vomiting, leak and port site problems .Long-term complications more than 1 month after surgery (e.g. nausea, vomiting, reflux, stricture, intestinal obstruction , hypoalbuminemia , anemia and calcium or iron or vitamin D , vitamin B12 deficiency and), excess weight loss and BMI were collected.

ELIGIBILITY:
Inclusion Criteria:Type 2 diabetic obese pateints -

Exclusion Criteria:patients age above 65 or below 18 years old, history of upper laparotomy, unfit for anesthesia or laparoscopy, major psychological instability and drug abuse.

-

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
excess weight loss | one year
  The percent of excess weight loss was calculated as follows: [(preoperative weight-follow up weight)/preoperative excess weight] ×100.
resolution of diabetes | one year
  Resolution of diabetes was defined in this study as a fasting plasma glucose level < 110 mg/dL or HbA1C level < 6 % without hypoglycemic medication at 1 year after surgery. whereas improvement was defined as a reduction of at least 25% in the fasting plasma glucose level and of at least 1% in the hemoglobin A1c level with hypoglycemic drug treatment

IPD SHARING:
Plan to Share IPD: Undecided